CLINICAL TRIAL: NCT05679037
Title: The Possible Role of Alpha-Lipoic Acid in Improving Endothelial Dysfunction and Atherosclerosis in Children With Type 1 Diabetes Mellitus
Brief Title: Role of Alpha-lipoic Acid in Diabetes Melitus Type 1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sara Ahmed mohamed Attia Harby, Administrator at faculty of pharmacy, Tanta university, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Role of ALA in diabetes
Record Dates: First submitted 2022-12-21; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Diabetes MellitusType 1
MeSH Terms: interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group who received insulin only plus placebo tablets (Placebo Comparator): (Placebo group; n=22) which will receive insulin plus placebo tablets once daily for 6 months.
  Interventions: Other: Placebo
- ALA group who received Alpha lipoic acid plus insulin (Active Comparator): (alpha-lipoic acid group; n=22) which will receive insulin plus ALA 600mg once daily for 6 months.
  Interventions: Drug: Alpha Lipoic Acid 600 MG Oral Capsule

INTERVENTIONS:
Other: Placebo — Inactive capsules
  Arms: Placebo group who received insulin only plus placebo tablets
Drug: Alpha Lipoic Acid 600 MG Oral Capsule — Universal antioxidant
  Other Names: Thioctic acid
  Arms: ALA group who received Alpha lipoic acid plus insulin

SUMMARY:
This study aims at investigating the possible effect of alpha-lipoic acid on endothelial dysfunction and atherosclerosis in children with type 1 diabetes mellitus.

DETAILED DESCRIPTION:
Endothelial dysfunction and alterations in vascular structure are early indicators of future cardiovascular events. The atherosclerotic changes begin much earlier than the appearance of clinical disease. Endothelial dysfunction in diabetes may be the result of a combination of multiple stressors. In the patients with type 1 diabetes, a significant increase in the concentrations of endothelial markers was already observed at the early stages of the disease including vascular cell adhesion molecules (VCAM-1), intercellular adhesion molecules (sICAM-1), soluble E- selectin E (sE-Selektin), asymmetric dimethylarginine (ADMA), plasminogen activator inhibitor 1 (PAI-1) because their concentrations increase rapidly in states of cellular stress. Increased carotid intima-media thickness (CIMT) is a structural marker for early atherosclerosis that correlates with cardio-vascular risk factors.

Alpha -lipoic acid supplementation may have role in Improving Endothelial Dysfunction and early Atherosclerosis due to its oxidative and anti-inflammatory effect.

ELIGIBILITY:
Inclusion Criteria:

* Children with T1DM on insulin therapy ≥ 0.5 IU/kg/day.
* Age range between 12 and < 18 years old.
* Both sex.
* Duration of diabetes ≥ 3 years.
* Glycated hemoglobin of ≥ 7.5%
* Patients who are previously evaluated for endothelial dysfunction and atherosclerosis.

Exclusion Criteria:

* Clinical evidence of heart failure, coronary artery disease, systemic hypertension, rheumatic fever, cardiomyopathy.
* Concurrent use of any medication other than insulin known to affect cardiac function (such as digitalis, angiotensin converting enzyme inhibitor, or β-blocker, etc…).
* Concurrent use of hyperlipidemia agents (Statin, fibrate).
* Concurrent use of antioxidants as selenium, vitamin C, vitamin E, etc..
* Patients with inflammatory conditions.
* Patients with conditions predispose to oxidative stress (obesity, COPD, etc…).
* Patients with liver disease.
* Patients with thyroid disease.
* Patients with seizures.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
The change in carotid artery intima-media thickness (CIMT) | Baseline and 6 months
  Measurement of carotid intima-media thickness (CIMT) which is mainly used to assess subclinical atherosclerosias and its assessment is based on ultrasound transducer

SECONDARY OUTCOMES:
The change in serum level of hs-CRP | Baseline and 6 months
  High sensitivity C- reactive protein (hs-CRP) which will be assessed by ELISA.
The change in serum level (MDA) | Baseline and 6 months
  Malondialdehyde (MDA) which will be assessed by colorimetric method.
The change in the serum level of VCAM-1 | Baseline and 6 months
  Vascular cell adhesion molecule-1 (VCAM-1) a marker of endothelial dysfunction which will be assessed by ELISA.
The change in the serum level of Apelin | Baseline and 6 months
  Serum Apelin a marker of atherosclerosis which will be assessed by ELISA
Lipid profile measuremt | Baseline and 6 months
  Total cholesterol (TC), triglyceride (TG) and HDL-C will be assessed by enzymatic colorimetric method.
Change in plasma level of (HbA1c %) | Baseline and 3,6 months
  Glycated hemoglobin (HbA1c %) will be measured by ion exchange micro-column chromatographic method.
Fast blood glucose measuremt | Baseline and 6 months
  Fasting blood glucose will be determined by glucose oxidase method.